CLINICAL TRIAL: NCT03220178
Title: PRECYCLE: Multicenter, Randomized Phase IV Intergroup Trial to Evaluate the Impact of eHealth-based Patient Reported Outcome (PRO) Assessment on Quality of Life in Patients With Hormone Receptor Positive, HER2 Negative Locally Advanced or Metastatic Breast Cancer Treated With Palbociclib and an Aromatase Inhibitor- or Palbociclib and Fulvestrant
Brief Title: Impact of eHealth-support on Quality of Life in Metastatic Breast Cancer Patients Treated With Palbociclib and Endocrine Therapy
Acronym: PRECYCLE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to COVID-19 pandemic, study cannot be finished in planned timeframe.
Sponsor: Palleos Healthcare GmbH (Industry)
Collaborators: WSG WOMEN´S HEALTHCARE STUDY GROUP (Unknown); Cankado GmbH (Industry); Pfizer (Industry); AGO-TraFo (Unknown); AGO-B (Unknown); Deutsche Gesellschaft für Hämatologie und Medizinische Onkologie e.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH001-PreCycle
Record Dates: First submitted 2017-07-06; First posted 2017-07-18 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Breast Neoplasm
Keywords: breast cancer; HER2 negative; hormone receptor positive; advanced; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — palbociclib; Fulvestrant; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CANKADO active (Experimental): CANKADO active is the fully functional CANKADO-based eHealth treatment support service, including a high density observation of patient reported outcome.
  Interventions: Drug: Palbociclib; Drug: Fulvestrant; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane
- CANKADO inform (Other): CANKADO inform stands for a CANKADO-based eHealth service with a personal login. For the patient , on-site surveys without feedback functions and a dosing tracker to document daily drug intake will be available. CANKADO inform will be used for the initial ePRO and further on-site ePROs. Patients can login from home, but they will only get text information about their disease and treatment. Further features will be unavailable.
  Interventions: Drug: Palbociclib; Drug: Fulvestrant; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane

INTERVENTIONS:
Drug: Palbociclib — Palbociclib 125mg/day orally dosed for 3 weeks followed by 1 week off; repeated for each treatment cycle
Drug: Fulvestrant — 500mg per use-after first application, again at wk2, then once per month
Drug: Anastrozole — 1mg per day
Drug: Letrozole — 2,5mg/day
Drug: Exemestane — 25mg/day

SUMMARY:
In this study the investigators assess the impact of the eHealth-supported therapy management system CANKADO on Quality of Life in patients with HR+, HER2-locally advanced or metastatic breast cancer treated with the cyclin dependent kinase 4/6 (CDK4/6) Inhibitor Palbociclib in combination with an aromatase inhibitor or fulvestrant. Furthermore this approach will be combined with biomarker screening to identify predictive markers for and to learn more about adherence, symptoms, response, and resistance.

DETAILED DESCRIPTION:
This is a multicenter (80 sites) , randomized, parallel-group, Phase IV clinical trial with the primary objective of testing the hypothesis of superiority for time to deterioration (TTD) in patients using the ePRO system CANKADO active over CANKADO inform version.

Eligible patients will have histologically or cytologically proven diagnosis of hormone receptor positive (HR+), human epidermal growth factor receptor 2 (HER2)- negative locally advanced or metastatic breast cancer and will be either candidates to receive palbociclib in combination with aromatase inhibitor or candidates to receive palbociclib in combination with fulvestrant for their locally advanced or metastatic disease. Patients who are candidates for palbociclib in combination with aromatase inhibitor (AI) or fulvestrant will not be candidates for curative therapies. For Patients who are candidates for palbociclib in combination with aromatase inhibitor or fulvestrant one prior line of chemotherapy for locally advanced or metastatic breast cancer is allowed in addition to a maximum of two lines of endocrine therapy. Patients will be stratified according their eligibility of receiving palbociclib with endocrine therapy (AI or fulvestrant) as first or later lines.

Patients allocated to the combination of palbociclib with aromatase inhibitor will receive:

* Palbociclib, 125 mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment and
* Aromatase inhibitor, orally once-daily (continuously).
* Pre- or peri-menopausal patients should additionally receive a Gonadotropin-Releasing-Hormon (GnRH)-agonist

Patients allocated to the combination of palbociclib with fulvestrant will receive:

* Palbociclib, 125 mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment and
* Fulvestrant , 500 mg, intramuscularly on Days 1 and 14 of Cycle 1, every 28 days (± 7 days) thereafter starting.
* Pre- or peri-menopausal patients should additionally receive a Gonadotropin-Releasing-Hormon (GnRH)-agonist

Patients of each treatment group (palbociclib / aromatase inhibitor and palbociclib/fulvestrant) will randomized 2:1 in the Intervention Arm A CANKADO active is the fully functional CANKADO-based eHealth treatment support service, including a high density observation of patient reported outcome (HDOB-PRO).

And in the Control Arm B CANKADO inform stands for a CANKADO-based eHealth service with a personal login. On-site surveys without feedback functions for the patient will be available. CANKADO inform will be used for the initial ePRO and further on-site ePROs. Patients can login from at home and can document their drug intake. Further features will not be available.

Patients will continue to receive study treatment together with the assigned ePRO assessment until investigator assessed disease progression, symptomatic deterioration, unacceptable toxicity, death, or withdrawal of consent, whichever occurs first. In addition, should palbociclib related toxicity mandate discontinuation; patients can continue to receive fulvestrant alone.

Patients discontinuing the active treatment phase will enter a follow-up period phase during survival further progression and new anti-cancer therapy information will be collected once a year up to 48 month after randomization.

In addition biomarkers will be assessed as a scientific program within this study. Tumor material (tumor tissue and Blood samples (plasma and serum)) will be collected. Tumor tissue from available primary tumor and available biopsies from recurrent disease will be collected. Blood samples will be collected at four time points (cycle 1 (C1D1), after 2 weeks (C1D14), after 12 weeks (C4D1), and upon progression (End of treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Post- or pre/peri-menopausal female patients, age ≥18 years
2. Patients with metastatic or locally advanced (non-operable) breast cancer disease
3. Patients who are appropriate candidates for aromatase inhibitor + palbociclib combination therapy OR Patients having already received endocrine therapy who are appropriate candidates for fulvestrant+ palbociclib combination therapy
4. Patient has not received treatment for locally advanced or metastatic disease OR Patient has received one prior line of chemotherapy and/or a maximum of two endocrine therapy lines for locally advanced or metastatic disease
5. Peri-/pre-menopausal patients should additionally receive a GnRH-agonist..
6. The tumor must be hormone-receptor positive
7. The tumor must be HER2-negative defined as either HER2 immunohistochemistry Score 0 or 1+ or as HER2-negative by in situ hybridization..
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
9. Adequate organ and marrow function before palbociclib treatment starts on C1D.
10. In case of patients of child bearing potential: negative pregnancy test (urine or serum) at baseline. Patients must agree to use highly effective non-hormonal contraception
11. Resolution of all acute toxic effects of prior therapy, including radiotherapy grade <1 (except toxicities not considered a safety risk for the patient) and recovery from surgical procedures
12. Signed Written Informed Consent
13. Willingness and capability to use CANKADO
14. Availability of hardware: Computer and/or tablet and/or smartphone with internet access

Exclusion Criteria:

1. Known hypersensitivity to aromatase inhibitor, fulvestrant, palbociclib or any of its excipients
2. Contraindication for aromatase inhibitor, fulvestrant or palbociclib; or GnRH-agonists (if pre-menopausal)
3. Prior treatment with any inhibitor of cyclin dependent kinase (CDK).
4. Patients with locally advanced or metastatic, symptomatic, visceral spread, who are at risk of life threatening complications in the short term
5. Known active uncontrolled or symptomatic central nervous system metastases
6. Current use of food or drugs known to be potent inhibitors or inducers of Cytochrome P450 3A4 (CYP3A4)
7. High cardiovascular risk, including, but not limited to recent myocardial infarction, severe/unstable angina, or severe cardiac dysrhythmias in the past 6 months of enrollment
8. Diagnosis of any second malignancy within the last 5 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix
9. Participation in other clinical trials involving investigational drug(s) (Phases 1-4) within 2 weeks before the current study begins and/or during study participation
10. Lactating women
11. Life expectancy < 3 months
12. Known infection with HIV, hepatitis B virus, or hepatitis C virus
13. Concurrent severe, uncontrolled systemic disease, social or psychiatric condition that might interfere with the planned treatment and with the patient's adherence to the protocol
14. Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
DQoL | From start of study treatment up to 4 years
  The event "deterioration of quality of life" (DQoL) will be measured every 28 days after enrolment using the FACT-B scale.

SECONDARY OUTCOMES:
Progression-free survival | From start of study treatment up to 4 years
  Progression-free survival (PFS) is considered to be the main clinical outcome and is defined as the time between treatment allocation and either first documentation of objective progression of disease (PD), as assessed by Investigator or death due to any cause in absence of PD.
Overall survival | From start of study treatment up to 4 years
  Overall survival (OS) is defined as the time between treatment allocation and death due to any cause.
Drug intake | From start of study treatment up to 4 years
  Daily electronic documentation of dosage and time of drug intake.
Global health status | From start of study treatment up to 4 years
  Daily electronic rating of overall health-related quality of life on a visual analogue scale (EQ-VAS) between 100 (best health imaginable) and 0 (worst health imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Iris Reiser, PhD, Study Director — Palleos Healthcare GmbH
Locations (1):
- University Hospital Mainz, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acquadro C, Berzon R, Dubois D, Leidy NK, Marquis P, Revicki D, Rothman M; PRO Harmonization Group. Incorporating the patient's perspective into drug development and communication: an ad hoc task force report of the Patient-Reported Outcomes (PRO) Harmonization Group meeting at the Food and Drug Administration, February 16, 2001. Value Health. 2003 Sep-Oct;6(5):522-31. doi: 10.1046/j.1524-4733.2003.65309.x. PMID 14627058
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Cella D, Hahn EA, Dineen K. Meaningful change in cancer-specific quality of life scores: differences between improvement and worsening. Qual Life Res. 2002 May;11(3):207-21. doi: 10.1023/a:1015276414526. PMID 12074259
- [Background] Cobos B, Haskard-Zolnierek K, Howard K. White coat hypertension: improving the patient-health care practitioner relationship. Psychol Res Behav Manag. 2015 May 2;8:133-41. doi: 10.2147/PRBM.S61192. eCollection 2015. PMID 25999772
- [Background] Coons SJ, Gwaltney CJ, Hays RD, Lundy JJ, Sloan JA, Revicki DA, Lenderking WR, Cella D, Basch E; ISPOR ePRO Task Force. Recommendations on evidence needed to support measurement equivalence between electronic and paper-based patient-reported outcome (PRO) measures: ISPOR ePRO Good Research Practices Task Force report. Value Health. 2009 Jun;12(4):419-29. doi: 10.1111/j.1524-4733.2008.00470.x. Epub 2008 Nov 11. PMID 19900250
- [Background] de Rond ME, de Wit R, van Dam FS, Muller MJ. A pain monitoring program for nurses: effects on communication, assessment and documentation of patients' pain. J Pain Symptom Manage. 2000 Dec;20(6):424-39. doi: 10.1016/s0885-3924(00)00209-8. PMID 11131261
- [Background] Deshpande PR, Rajan S, Sudeepthi BL, Abdul Nazir CP. Patient-reported outcomes: A new era in clinical research. Perspect Clin Res. 2011 Oct;2(4):137-44. doi: 10.4103/2229-3485.86879. PMID 22145124
- [Background] Detmar SB, Muller MJ, Schornagel JH, Wever LD, Aaronson NK. Health-related quality-of-life assessments and patient-physician communication: a randomized controlled trial. JAMA. 2002 Dec 18;288(23):3027-34. doi: 10.1001/jama.288.23.3027. PMID 12479768
- [Background] Dorand RD, Nthale J, Myers JT, Barkauskas DS, Avril S, Chirieleison SM, Pareek TK, Abbott DW, Stearns DS, Letterio JJ, Huang AY, Petrosiute A. Cdk5 disruption attenuates tumor PD-L1 expression and promotes antitumor immunity. Science. 2016 Jul 22;353(6297):399-403. doi: 10.1126/science.aae0477. Epub 2016 Jul 21. PMID 27463676
- [Background] Eton DT, Cella D, Yost KJ, Yount SE, Peterman AH, Neuberg DS, Sledge GW, Wood WC. A combination of distribution- and anchor-based approaches determined minimally important differences (MIDs) for four endpoints in a breast cancer scale. J Clin Epidemiol. 2004 Sep;57(9):898-910. doi: 10.1016/j.jclinepi.2004.01.012. PMID 15504633
- [Background] Finn RS, Crown JP, Lang I, Boer K, Bondarenko IM, Kulyk SO, Ettl J, Patel R, Pinter T, Schmidt M, Shparyk Y, Thummala AR, Voytko NL, Fowst C, Huang X, Kim ST, Randolph S, Slamon DJ. The cyclin-dependent kinase 4/6 inhibitor palbociclib in combination with letrozole versus letrozole alone as first-line treatment of oestrogen receptor-positive, HER2-negative, advanced breast cancer (PALOMA-1/TRIO-18): a randomised phase 2 study. Lancet Oncol. 2015 Jan;16(1):25-35. doi: 10.1016/S1470-2045(14)71159-3. Epub 2014 Dec 16. PMID 25524798
- [Background] Finn RS, Martin M, Rugo HS, Jones SE, Im SA, Gelmon KA, Harbeck N, Lipatov ON, Walshe JM, Moulder SL, Gauthier ER, Lu D, Randolph S, Diéras V, Slamon DJ. PALOMA-2: Primary results from a phase III trial of palbociclib (P) with letrozole (L) compared with letrozole alone in post-menopausal women with ER+/HER2- advanced breast cancer (ABC). J Clin Oncol 34, 2016 (suppl; abstr 507)
- [Background] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- [Background] Harbeck, N., R. Wuerstlein and T. Schinkoethe (2015).
- [Background] U.S. Department of Health and Human Services FDA Center for Drug Evaluation and Research; U.S. Department of Health and Human Services FDA Center for Biologics Evaluation and Research; U.S. Department of Health and Human Services FDA Center for Devices and Radiological Health. Guidance for industry: patient-reported outcome measures: use in medical product development to support labeling claims: draft guidance. Health Qual Life Outcomes. 2006 Oct 11;4:79. doi: 10.1186/1477-7525-4-79. PMID 17034633
- [Background] Kalbfleisch, J.D., Prentice, R. L. (2002). "The statistical analysis of failure time data" (2nd Ed.) John Wily & Sons, p. 224
- [Background] Miller RD, Walsh TD. Psychosocial aspects of palliative care in advanced cancer. J Pain Symptom Manage. 1991 Jan;6(1):24-9. doi: 10.1016/0885-3924(91)90068-f. PMID 1703198
- [Background] Pickering TG, James GD, Boddie C, Harshfield GA, Blank S, Laragh JH. How common is white coat hypertension? JAMA. 1988 Jan 8;259(2):225-8. PMID 3336140
- [Background] Politi MC, Clark MA, Ombao H, Dizon D, Elwyn G. Communicating uncertainty can lead to less decision satisfaction: a necessary cost of involving patients in shared decision making? Health Expect. 2011 Mar;14(1):84-91. doi: 10.1111/j.1369-7625.2010.00626.x. Epub 2010 Sep 23. PMID 20860780
- [Background] Rosenbloom DI, Hill AL, Rabi SA, Siliciano RF, Nowak MA. Antiretroviral dynamics determines HIV evolution and predicts therapy outcome. Nat Med. 2012 Sep;18(9):1378-85. doi: 10.1038/nm.2892. PMID 22941277
- [Background] Schoenfeld, D. A., Tsiatis, A. A. (1987)."A modified log rank test for highly stratified data." Biometrika, 167-175
- [Background] Townsend A, Leese J, Adam P, McDonald M, Li LC, Kerr S, Backman CL. eHealth, Participatory Medicine, and Ethical Care: A Focus Group Study of Patients' and Health Care Providers' Use of Health-Related Internet Information. J Med Internet Res. 2015 Jun 22;17(6):e155. doi: 10.2196/jmir.3792. PMID 26099267
- [Background] Turner NC, Ro J, Andre F, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Huang Bartlett C, Zhang K, Giorgetti C, Randolph S, Koehler M, Cristofanilli M; PALOMA3 Study Group. Palbociclib in Hormone-Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2015 Jul 16;373(3):209-19. doi: 10.1056/NEJMoa1505270. Epub 2015 Jun 1. PMID 26030518
- [Background] Vanden Bush TJ, Bishop GA. CDK-mediated regulation of cell functions via c-Jun phosphorylation and AP-1 activation. PLoS One. 2011 Apr 29;6(4):e19468. doi: 10.1371/journal.pone.0019468. PMID 21559334
- [Background] Wells AD, Morawski PA. New roles for cyclin-dependent kinases in T cell biology: linking cell division and differentiation. Nat Rev Immunol. 2014 Apr;14(4):261-70. doi: 10.1038/nri3625. Epub 2014 Mar 7. PMID 24603166
- [Background] Yost KJ, Eton DT. Combining distribution- and anchor-based approaches to determine minimally important differences: the FACIT experience. Eval Health Prof. 2005 Jun;28(2):172-91. doi: 10.1177/0163278705275340. PMID 15851772
- [Derived] Harbeck N, Fasching PA, Wuerstlein R, Degenhardt T, Luftner D, Kates RE, Schumacher J, Rath P, Hoffmann O, Lorenz R, Decker T, Reinisch M, Gohler T, Staib P, Gluz O, Schinkothe T, Schmidt M; AGO-B WSG PreCycle investigators (see Appendix 1). Significantly longer time to deterioration of quality of life due to CANKADO PRO-React eHealth support in HR+ HER2- metastatic breast cancer patients receiving palbociclib and endocrine therapy: primary outcome analysis of the multicenter randomized AGO-B WSG PreCycle trial. Ann Oncol. 2023 Aug;34(8):660-669. doi: 10.1016/j.annonc.2023.05.003. Epub 2023 May 16. PMID 37201751